CLINICAL TRIAL: NCT00192894
Title: Cardiac Output Changes During Onset of Spinal Anesthesia in Elderly Patients
Brief Title: New Methods to Detect a Decrease in Heart Function
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Danish Medical Research Council (Other); Oberstinde Kirsten Jensa la Cours Foundation (Other)
Responsible Party: Principal Investigator, Lars S. Rasmussen, MD, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: 22-04-0019
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Orthopedic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study was to evaluate the changes in heart function during onset of spinal anesthesia using a new and less invasive method, the LidcoTMplus.

DETAILED DESCRIPTION:
The incidence of hypotension during onset of spinal anesthesia in elderly patients varies from 27% to 80% depending on which definition being used. Studies of cardiac output (CO) has shown that it is maintained or only slightly decreased .

Unfortunately, the time-resolution in these studies is often several minutes, and the description of changes is consequently often a start-to-end relation rather than a description of the dynamic changes during onset of spinal anesthesia.

A recent advance in measuring CO is the LiDCOTMplus hemodynamic monitor, which has proved reliable compared to pulmonary artery catheters in various intensive care settings. This monitor allows for beat-to-beat measuring during various procedures and thus early warning of hemodynamic events.

Another method with potential for early warning of decreased perfusion is near-infrared spectroscopy (NIRS). NIRS is used for continuous and non-invasive monitoring of cerebral oxygen saturation (ScO2) and even a small reduction has recently shown to predict maternal hypotension during caesarian section.

The aim of our study was to describe the changes in CO during onset of spinal anesthesia in elderly patients using a method with high time-resolution. We also attempted to evaluate NIRS as predictor of hemodynamic events.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Elective orthopedic or plastic lower limp surgery
* in spinal anesthesia

Exclusion Criteria:

* Body weight <40 kg
* Currently in treatment with lithium
* Evidence of aortic valve regurgitation

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients undergoing spinal anaesthesia
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2004-05-15 (Actual); Primary Completion 2005-03-15 (Actual); Study Completion 2005-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars S. Rasmussen, MD, PhD, Study Chair — Department of anaesthesia, 4231, Center of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Department of anaesthesia, 4231, Center of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark